CLINICAL TRIAL: NCT07295392
Title: Serum Uromodulin Prognostic Value in Sepsis Induced AKI
Brief Title: Is There Any Prognostic Value of Serum Uromodulin in Sepsis Induced AKI.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaymaa Ibrahim Mohammed Hassan, Resistant doctor in internal medicine department at Assiut university, Assiut University
Other Study IDs: Uromodulin in AKI
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Acute Kidney Injury
Keywords: Serum uromodulin
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine whether baseline (day 0; day of diagnosis),day 7 and on discharge serum uromodulin levels help predict clinical outcomes in adult patients with sepsis induced AKI.

DETAILED DESCRIPTION:
Sepsis remains a leading cause of morbidity and mortality worldwide, with risk rising as organs failure accumulate, particularly when acute kidney injury (AKI) develops. AKI complicates nearly half of all septic episodes in ICU and is independently associated with poorer short- and long-term outcomes. Current prognostic tools as SOFA score , serum creatinine, urine output, NGAL and KIM-1have limited prognostic value. They often detect injury only after significant damage has occurred.

Uromodulin, the most abundant urinary protein produced by the renal thick ascending limb, is present in small amounts in the circulation. Experimental models reveal that uromodulin deficiency worsens sepsis outcomes, while administration of exogenous uromodulin can reduce mortality . In clinical studies of septic patients, early rises in circulating uromodulin are observed, yet those who go on to develop AKI or die tend to have lower levels at presentation. Genetic analyses, however, have not definitively proven a causal protective role for baseline uromodulin.

It has roles in tubular protection, immune modulation, and infection control, These important physiological functions may translate into valuable prognostic tools that may aid in predicting clinical outcomes. Serum uromodulin may serve as an early indicator of both renal tubular integrity and host defence capacity-qualities not captured by existing markers. Assessing serum uromodulin at time of diagnosis(day 0), day 7 and at time of discharge may predict recovery or progression of AKI. Establishing the prognostic value of uromodulin could enable early risk stratification, guide tailored interventions, and inform clinical decision-making, potentially improving outcomes in sepsis-induced AKI.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Septic patients with AKI: Diagnosis of sepsis is based on combination of variables including Sepsis-3 criteria within 24 hours of ICU admission(suspected or confirmed infection on clinical , lab and imaging evidence , acute increase in SOFA score =>2 points( or presence of septic shock). The latter is defined by a vasopressor requirement to maintain a mean arterial pressure of 65 mm Hg or greater and serum lactate level greater than 2 mmol/L (>18 mg/dL) in the absence of hypovolemia (Singer et al 2016).
3. Diagnosis of AKI according to KDIGO-criteria ( increase creatinine by =>0.3 mg/dl ( =>26.5 micmol/l ) within 48 hrs or increase cr =>1.5 × baseline within 7days or urine output < 0.5 ml / kg / hr for => 6hrs)
4. Informed consent obtained and in case patient is unable to sign the consent his next of kin or has power

Exclusion Criteria:

1. Patients diagnosed with ESRD or kidney transplantation
2. Other causes of AKI
3. Pregnancy related causes of AKI
4. Active immunosuppressive therapy (e.g., high-dose steroids, chemotherapy)
5. Patients with background of adult polycystic kidney disease
6. Patients with cardiac failure
7. Patients with solitary kidney because of small renal mass that could affect uromodulin level.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who is recently diagnosed with AKI due to sepsis meeting the previously mentioned criteria and doesn't have the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-03-10 (Estimated); Primary Completion 2026-12-10 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Serum Uromodulin as a Predictor of Acute Kidney Injury Outcome in Septic Patients | 30 days
  To assess whether serum uromodulin levels measured at ICU admission (day 0), day 7, and at ICU discharge can predict AKI outcome (complete renal recovery versus progression to chronic kidney disease), length of ICU stay, and 30-day all-cause mortality in adult patients with sepsis-induced acute kidney injury.

SECONDARY OUTCOMES:
2.1.Correlation Between Serum Uromodulin Levels and Need for Renal Replacement Therapy. 2.2.Correlation Between Serum Uromodulin Levels and SOFA Score. 2.3.Correlation Between Serum Uromodulin Levels and AKI Severity. | From ICU admission to ICU discharge.